CLINICAL TRIAL: NCT03678987
Title: Mycophenolate Mofetil in Systemic Sclerosis: A Phase 1 Pharmacokinetic Study of Orally Ingested Mycophenolate Mofetil Tablets in Patients Suffering From Systemic Sclerosis
Brief Title: Mycophenolate Mofetil Pharmacokinetics in Systemic Sclerosis
Acronym: MMFSSC
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Kristofer Andreasson, Principal Investigator, Region Skane
Other Study IDs: 2018-002105-54
Record Dates: First submitted 2018-09-13; First posted 2018-09-20 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Systemic Sclerosis; Gastrointestinal Complication
Keywords: pharmacokinetics; mycophenolate mofetil
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SSc on MMF: Patients with systemic sclerosis using mycophenolate mofetil (mycophenolic acid, MMF) since >3 months.
  During a 6 hour time period, P-MPA concentration will be measured 4 times.
  Interventions: Diagnostic Test: P-MPA concentration; Drug: mycophenolic acid

INTERVENTIONS:
Diagnostic Test: P-MPA concentration — We will calculate AUC_0-12 of MPA based on 4 measurements of P-MPA
Drug: mycophenolic acid — Patient will ingest mycophenolic acid as prescribed by their physician under the surveillance of an investigator.
  Other Names: cellcept; mycophenolate mofetil

SUMMARY:
Drug of investigation: Mycophenolate mofetil (MMF), given orally as a tablet twice daily.

Dosage of drug: This study recruits patients who have been prescribed a steady dose of MMF in the range between 1000 and 3000 mg daily by their physician.

Design: This is an open-label PK study.

Disease studied: Systemic sclerosis (SSC, scleroderma).

Variables assessed: Estimated AUC0-12 for MMF. Gastrointestinal manifestations of SSc. Concomitant medication.

Study population:

Inclusion criteria: Diagnosis of SSC fulfilling the 2013 classification criteria for this disease. Participant should have been prescribed a stable dose of MMF tablets, taken twice daily, for at least 3 months prior to the study.

Exclusion criteria: Failure to comply with study protocol. Limited access to repeated venous puncture. Recipient of organ transplant. Pulmonary arterial hypertension.

Number of participants: The study aims at the inclusion of 35 subjects.

Primary objective: To investigate the PK of orally ingested MMF in SSC.

Secondary objectives:

1. To investigate how SSC manifested in the gastrointestinal (GI) tract may alter the PK of MMF.
2. To investigate how the PK of MMF in SSc is altered by medications often used in SSC, i.e. proton pump inhibitors (PPI), NSAID and calcium channel blockers.

DETAILED DESCRIPTION:
DESIGN AND ASSESSMENT SCHEDULE Study participants will take their medication, including the study drug, as prescribed by their ordinary physician. Study participant will note what they had for breakfast.

The study-timespan for the individual study participant is estimated to maximum 8 hours.

Blood samples will be drawn from a subcutaneous venous port if available. If not available, subjects will be receive a peripheral venous catheter that is to be used for repeated blood sampling. If usage of such a catheter fails during the study day, blood samples will be drawn from repeated venipunctures.

VARIABLES STUDIED

The following variables will be studied:

Plasma-MMF-concentration: Will be measured by approved laboratory, Skåne UniversityHospital, using high performance liquid chromatography. AUC 0_12 will be calculated as suggested by de Winter, Neumann, van Hest et. al., Ther Drug Mon 2009;31(3):382-390.

Kidney and liver function: Serum samples will be analysed regarding kidney function and eGFR will be calculated from creatinin and cystatin C. Liver function will be assessed by AST, ALT, GT and ALP. Hematological characteristics will be noted.

GI manifestations of SSc: Fecal calprotectin, will be assayed by ELISA (Calpro, Lysaker, Norway) at University Hospital Lund. Malnutrition will evaluated in reference to the validated Malnutrition Universal Screening Tool (MUST). S-transthyretin, vitamin B12, folic acid, iron and zink and S-albumin will be assessed as markers of malnutrition. The intestinal flora will be assessed by microbiological analysis of fecal sampling (Genetic Analysis AS, Oslo, Norway).

Pregnancy: Will be evaluated by urine test.

Questionnaire: Regarding concomitant medication and the UCLA SCTC GIT 2.0 (Swedish version) will be given to each study participant.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of SSC according to the 2013 ACR/EULAR classification criteria
* above 18 years of age
* fluent in Swedish and able to understand the study protocol and "Patient information"
* being prescribed and using a fixed dos (1000-3000 mg daily) of MMF tablet, Cellcept or substitutable medical product, twice daily since at least 3 months
* the study participant's written and informed consent
* women in child-bearing age should use contraception

Exclusion Criteria:

* Recipient of a solid organ transplant
* Pregnancy or lactation
* The presence of renal failure (defined as eGFR < 30 ml/min)
* A history of complicated venipunctures defined as
* a history of any venipuncture within the last year that required three or more attempts in order to succeed or
* a decision has been made that the patient should receive a subcutaneous venous port because of complicated venipunctures.

If the patient has a functioning subcutaneous venous port, the above criteria does not apply if venous sampling has been uncomplicated from this port.

* A history of hypersensitivity reactions to MMF
* Patients diagnosed with any kind of acute infection during the one (1) week preceding the study day
* A history of gastrointestinal surgery that includes resection of any port of the ventricle, small intestine, large intestine or liver (except for surgery for appendicitis, gall bladder resection or hemorrhoids, which do not constitute reasons for exclusion)
* Pulmonary arterial hypertension
* Anemia, defined as Hb < 100 g/L during the last 4 weeks The patient will be informed about the study and sign informed consent before study commences.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis using a stable dose of mycophenolate mofetil.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Individual plasma concentrations of mycophenolic acid | 1 day
  By 4 measurements of P-MPA during a 6 hour time period we will estimate the individual drug exposition expressed as Area Under the Curve (AUC) 0-12 for this medicine and calculated as suggested by Abd Rahman 2014 (reference 3).

SECONDARY OUTCOMES:
Correlation between F-calprotectin and the AUC of P-MPA | 1 day
  To investigate how gastrointestinal inflammation as measured by F-calprotectin correlate with the AUC of P-MPA
Correlation between the USCLA SCTC GIT-2.0 questionnaire and the AUC of P-MPA | 1 day
  To investigate how the gastrointestinal manifestations of SSc, assessed by a SSc-specific questionnaire, correlate with the AUC of P-MPA
Correlation between the Malnutrition Universal Screening Tool (MUST) and the AUC of P-MPA | 1 day
  To investigate if malnutrition, assessed by the MUST, correlate with the AUC of P-MPA
Correlation between the precense of dysbiosis, as defined by the GA-MAP Dysbiosis Test and the AUC of P-MPA | 1 day
  To investigate if intestinal dysbiosis, assessed by the a validated test available through Genetic Analysis, Oslo Norway, is associated with the AUC of P-MPA
Association between the AUC of P-MPA and the concomitant medication with a) NSAID, b) proton-pump inhibitors and c) Ca-channel blockers | 1 day
  To compare the AUC of P-MPA in patients with and without the above mentionened concomitant medication

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer Andréasson, MD PhD, Principal Investigator — Region Skane
Locations (1):
- Reumatologi SUS Lund, Region Skåne, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This issue will be discussed with the Ethical board.

REFERENCES:
- [Background] Volkmann ER, Tashkin DP, Li N, Roth MD, Khanna D, Hoffmann-Vold AM, Kim G, Goldin J, Clements PJ, Furst DE, Elashoff RM. Mycophenolate Mofetil Versus Placebo for Systemic Sclerosis-Related Interstitial Lung Disease: An Analysis of Scleroderma Lung Studies I and II. Arthritis Rheumatol. 2017 Jul;69(7):1451-1460. doi: 10.1002/art.40114. Epub 2017 May 23. PMID 28376288
- [Background] McCune WJ, Al Abbas M. Mycophenolate mofetil, for rheumatic diseases: should we monitor the area under the curve? Curr Opin Rheumatol. 2018 May;30(3):229-230. doi: 10.1097/BOR.0000000000000501. No abstract available. PMID 29538009
- [Background] Abd Rahman AN, Tett SE, Staatz CE. How accurate and precise are limited sampling strategies in estimating exposure to mycophenolic acid in people with autoimmune disease? Clin Pharmacokinet. 2014 Mar;53(3):227-245. doi: 10.1007/s40262-013-0124-z. PMID 24327238
- [Background] de Winter BC, Neumann I, van Hest RM, van Gelder T, Mathot RA. Limited sampling strategies for therapeutic drug monitoring of mycophenolate mofetil therapy in patients with autoimmune disease. Ther Drug Monit. 2009 Jun;31(3):382-90. doi: 10.1097/FTD.0b013e3181a23f1a. PMID 19363460